CLINICAL TRIAL: NCT05614882
Title: New Model of Stroke Education
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000033911
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Individuals in this study will be based from a convenience sample from the Rehabilitation and Wellness Center in Milford, Connecticut. Participants will be admitted post-stroke after being diagnosed with stroke of mild to moderate severity. Individuals will be over 18 years of age with no history of prior stroke who are able to read basic information, having no more than a mild aphasia with intact language comprehension skills who speak English or Spanish (assessment materials are available in these two languages).
  All the participants will receive a health literacy assessment and based on their scores will be categorized into a high health literacy (HHL) or low health literacy group (LHL) prior to randomization. Anticipated enrollment of 20 for pilot and 200 for larger study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written Stroke Education (Active Comparator): Participants in this arm will be given the current written standard of care for stroke education. Assessments will be completed during the participants inpatient stay.
  Interventions: Behavioral: Written Stroke Education
- Verbal Stroke Education (Experimental): Participants in this arm will be given the experimental verbal stroke education. Assessments will be completed during the participants inpatient stay.
  Interventions: Behavioral: Verbal Stroke Education

INTERVENTIONS:
Behavioral: Written Stroke Education — The written education will be provided in the stroke folder currently in use by the Yale New Haven Health system. This written information is presented in a stroke folder and includes how to respond to the signs of stroke, dialing 9-1-1, following up with a health care provider after hospitalization due to a stroke and the importance of medication management as well as stroke risk factors, healthy eating habits, exercise habits, common changes following a stroke, stroke recurrence and stroke types. After being given two days to review the materials, patients will be asked to complete the stroke knowledge test (SKT). All participants will receive a health literacy assessment and based on their scores will be categorized into a high health literacy (HHL) or low health literacy group (LHL) prior to randomization.
  Arms: Written Stroke Education
Behavioral: Verbal Stroke Education — Participants in the verbal education group will be provided with education over two days from therapists including occupational therapy, physical therapy, speech therapy as well as a physician or nurse. The disciplines will present general stroke information including causes, risk factors, prevention, nutrition and exercise recommendations, importance of managing chronic conditions and the significance of medication compliance. After the verbal education topics are presented, the participants will be tested with the stroke knowledge test (SKT) to measure learning. All the participants will receive a health literacy assessment and based on their scores will be categorized into a high health literacy (HHL) or low health literacy group (LHL) prior to randomization.
  Arms: Verbal Stroke Education

SUMMARY:
The main goal of this study is to reorganize how stroke educational materials are given to patients from written delivery of information to using verbal delivery of information. Another goal is to compare post stroke behavior and medication compliance in participants receiving the new verbal model of stroke education vs. those receiving the current written stroke education.

The main question[s] it aims to answer are:

* Does the current delivery of stroke education provide the necessary knowledge base for patients who have suffered a stroke as measured by a stroke questionnaire?
* Does verbal education provide better understanding for patients post-stroke?
* Are patients more likely to be compliant with medications and followup visits with their medical team after receiving verbal education? Participants will receive a health literacy assessment and based on their scores will be categorized into a high health literacy (HHL) or low health literacy group (LHL). Individuals in both literacy groups will be randomized into receiving verbal or written stroke education. All participants will be tested with the stroke knowledge assessment to measure learning after education.

Researchers will compare written to verbal education to see if verbal results in more stroke education and compliance.

DETAILED DESCRIPTION:
The primary objective of this study is to restructure the current model of stroke education using verbal delivery of information that is accessible and understood by individuals of different cultural backgrounds and various literacy levels. Participants in this study will be provided with a new model of stroke education through verbal communication to educate them on factors related to stroke using vocabulary that is more familiar and understood by individuals with lower literacy levels. The current delivery of stroke information is carried out through a model that involves mainly written communication. Data will be collected to better understand the efficacy of the current written model of stroke education compared to the new verbal education and determine which of the two methods of delivering information is more compatible with the literacy levels of the community served by Yale New Haven Hospital.

The second part of the study, participants' electronic medical record (EMR) will be reviewed at 1, 3, 6 and 12 months post stroke to evaluate the attendance post stroke follow up visits, post stroke blood pressure readings and overall medication compliance.

Participants in this study will be based from a convenience sample from the Rehabilitation and Wellness Center in Milford, Connecticut. Participants will be admitted post-stroke after being diagnosed with stroke of mild to moderate severity.

All the participants will receive a health literacy assessment and based on their scores will be categorized into a high health literacy (HHL) or low health literacy group (LHL) prior to randomization.

Assessments will be completed during the participants inpatient stay. A run in pilot study of 20 anticipated participants will be carried out prior to the larger study. The larger study was registered in anticipation of NIH funding.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age at time of stroke.
* Documentation of a stroke diagnosis as evidenced by one or more clinical features consistent with deficits in physical mobility, mild deficits in language

Exclusion Criteria:

* Documented history of stroke
* Documented cognitive deficits
* Individuals <18 years of age
* Individuals who are unable to provide consent
* Those who are pregnant will be excluded from this sample (pregnancy tests are typically completed on admission, for applicable individuals).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Stroke Knowledge Test (SKT) | 1 day post intervention
  SKT is a 20 question assessment to determine if written or verbal delivery of post stroke education was more successful in educating participants. The assessment is scored as a percentage of correct questions out of a total of 20 questions. Higher scores indicate more educated on stroke.

SECONDARY OUTCOMES:
Count of post stroke follow up visits attended | Month 1 up to Month 12 post discharge
  Electronic medical records will be reviewed at 1, 3, 6 and 12 months post discharge to evaluate if participants had post stroke follow up visits with their care providers (recorded as yes/no). This will demonstrate which method is more likely to support patients in gathering information that is needed to manage their chronic conditions, maintaining compliance and decrease their chance of stroke recurrence.
Count of post stroke blood pressure readings above 130/80 mmHG systolic | Month 1 up to Month 12 post discharge
  Electronic medical records will be reviewed at 1, 3, 6 and 12 months post discharge to monitor how many post stroke blood pressure readings are above 130/80 mmHG systolic.This will demonstrate which method is more likely to support patients in gathering information that is needed to manage their chronic conditions, maintaining compliance and decrease their chance of stroke recurrence.
Medical compliance measured by count of prescriptions filled | Month 1 up to Month 12 post discharge
  Electronic medical records will be reviewed at 1, 3, 6 and 12 months post discharge to count the number of prescriptions filled that were ordered by the provider. Medical compliance will be assessed by the number of prescriptions filled. This will demonstrate which method is more likely to support patients in gathering information that is needed to manage their chronic conditions, maintaining compliance and decrease their chance of stroke recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Necolle Morgado-Vega, MD, Principal Investigator — Yale University
Locations (1):
- YNHH Rehabilitation & Wellness Center, Milford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes